#### Official Title:

Using In-depth Interviews to Examine Neighborhood Influence on Parenting Practices Regarding Youth Outdoor Play and Physical Activity

NCT #: NA
Date Updated: 04/06/2017
Date Approved by IRB: 4/20/2017

# FOR AN ADULT INFORMED CONSENT - PART I

Using In-depth Interviews to Examine Neighborhood

Title of Study: Influence on Parenting Practices Regarding Youth

Outdoor Play and Physical Activity.

#### What you should know about a research study

 We give you this consent form so that you may read about the purpose, risks and benefits of this research study.

- The main goal of research studies is to gain knowledge that may help people in the future.
- You have the right to refuse to take part, or agree to take part now and change your mind later on.
- Please review this consent form carefully and ask any questions before you make a decision.
- Your participation is voluntary.
- By signing this consent form, you agree to participate in the study as it is described.

#### 1- Who is doing the study?

Investigator Information:

Principal Investigator: Maura Kepper, PhD

1-225-763-2698

Sub Investigators: Stephanie Broyles, PhD

Amanda Staiano, PhD Peter Katzmarzyk, PhD

Dr. Kepper leads this study. We expect 32 people to be enrolled in this study. The study will last 2 years, but you will only be in this study during this study visit. Your expected time in this study will be 1-2 hours.

#### 2- Where is the study being conducted?

This study takes place in private room located within Pennington Biomedical Research Center or at a private room in a community location (i.e. YMCA or EBPRL branch).

#### 3- What is the purpose of this study?

The purpose of this study is to use qualitative methods (in-depth interviews) among parents/guardians living in varied neighborhood environments (supportive and

Version Date: use current date Page 2 of 5

| #PBRC |
|-------|

unsupportive physical environments) to gain in-depth information and perspectives of the social environment's influence on constrained outdoor play practices. Furthermore, this study will identify how parents/guardians experience poor physical characteristics in their neighborhood and physical environmental characteristics influence perspectives shared during in-depth interviews.

#### 4- Who is eligible to participate in the study?

You may be eligible to participate in the study if:

Your child completed baseline measures for the TIGER Kids Study at PBRC.

#### You may not be eligible to participate in the study if:

- Your child did not complete baseline measures for the TIGER Kids Study at PBRC.
- You did not report a home address at the baseline TIGER Kids study visit.
- You are unwilling or unable to participate in an in-depth interview.

#### 5- What will happen to you if you take part in the study?

If you agree to join this study and sign this consent, we will ask you to complete a short confidential questionnaire describing some basic demographic information. Next, you will participate in 1-2 hour in-depth interview regarding your neighborhood environment, your parenting practices regarding your child's outdoor play and your child's physical activity behaviors. We will be audio-taping the interview to make sure we don't miss anything that you say. The researcher will ask you to use only first names during the interview. This will help us keep the audio-tape confidential and protect the privacy of you and anyone discussed.

#### 6- What are the possible risks and discomforts?

There are no foreseeable risks due to participation in this study. The interviews will not include any sensitive topics that could make participants uncomfortable. However, you do not have to answer any questions you do not want to answer.

#### 7- What are the possible benefits?

We cannot promise any benefits from your being in the study. The input you provide us during this interview will be used to identify community strategies to increase children's outdoor play and may inform future policy changes for neighborhood environments to promote health.

### 8- If you do not want to take part in the study, are there other choices?

You have the choice at any time not to participate in this research study. If you choose not to participate, any health benefits to which you are entitled will not be affected in any way.

| #PBRC |
|-------|
| #PBRC |

#### 9- If you have any questions or problems, whom can you call?

If you have any questions about your rights as a research volunteer, you should call the Institutional Review Board Office at 225-763-2693 or the Executive Director of Pennington Biomedical at 225-763-2513. If you have any questions about the research study, contact Maura Kepper at 1-225-763-2698.

#### 10- What information will be kept private?

Every effort will be made to maintain the confidentiality of your study records. However, someone from the National Institutes of Health, the Pennington Biomedical Research Center, and the Eunice Kennedy Shriver Nation Institute of Child Health and Human Development (NICHD) (the sponsor) may inspect and/or copy the medical records related to the study. Results of the study may be published; however, we will keep your name and other identifying information private. Other than as set forth above, your identity will remain confidential unless disclosure is required by law.

#### 11- Can your taking part in the study end early?

Dr. Maura Kepper can withdraw you from the study for any reason or for no reason. You may withdraw from the study at any time without penalty; however, all data Pennington Biomedical has previously collected cannot be removed from the study. Possible reasons for withdrawal include unwillingness on behalf of the participant to participate in the study or cooperate with study staff.

## 12- What if information becomes available that might affect your decision to stay in the study?

During the course of this study there may be new findings from this or other research which may affect your willingness to continue participation. Information concerning any such new findings will be provided to you.

### 13- What charges will you have to pay?

None.

#### 14- What payment will you receive?

If you agree to take part, we will pay you \$25 upon completion of the in-depth interview. Your check will be requested from the LSU payroll department when you complete the study. It usually takes about 3-4 weeks for it to arrive at Pennington Biomedical Research Center. The payment will then be mailed to your home address.

### 15- Will you be compensated for a study-related injury or medical illness?

No form of compensation for medical treatment or for other damages (i.e., lost wages, time lost from work, etc.) is available from the Pennington Biomedical Research Center. In the event of injury or medical illness resulting from the research procedures in which you participate, you will be referred to a treatment facility. Medical treatment may be provided at your expense or at the expense of your health care insurer (e.g., Medicare,

| #PBRC |
|---|
| Medicaid, Blue Cross-Blue Shield, Dental Insurer, etc.) which may or may not provide coverage. The Pennington Biomedical Research Center is a research facility and provides medical treatment only as part of research protocols. Should you require ongoing medical treatments, they must be provided by community physicians and hospitals. |
| <b>16- Signatures</b> The study has been discussed with me and all my questions have been answered. I understand that additional questions regarding the study should be directed to the study investigators. I agree with the terms above and acknowledge that I will be given a copy of this signed consent form. |
| With my signature, I also acknowledge that I have been given either today or in the past a copy of the Notice of Privacy Practices for Protected Health Information. |
| Printed Name of Volunteer |
| Signature of Volunteer Date |
| Printed Name of Person Administering Informed Consent |

<u>Dr. Maura Kepper</u> Principal Investigator

Signature of Person Administering Informed Consent

Date